CLINICAL TRIAL: NCT01757223
Title: Phase I/II Study, Administration of AdVEGF-All6A+, a Replication Deficient Adenovirus Vector Expressing a cDNA/Genomic Hybrid of Human Vascular Endothelial Growth Factor to the Ischemic Myocardium...
Brief Title: Administration of AdVEGF-All6A+ to Myocardium of Individuals With Diffuse CAD Via Minimally Invasive Surgery
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closure due to lack of funding.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1204012330; 1201-1145 (Other: Recombinant DNA Advisory Commitee)
Record Dates: First submitted 2012-10-10; First posted 2012-12-28 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Diffuse Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A, Group 1 - 10^8 pu (Experimental): Part A is a dose-escalation, open-label study, administering 3 doses of AdVEGF-All6A+ to n=9 individuals, with n=3 each at 10^8, 10^9, and 10^10 particle units. The purpose of Part A is to determine the highest tolerable dose. Group 1 will receive 10^8 particle units.
  Interventions: Biological: AdVEGF-All6A+
- Part A, Group 2 - 10^9 pu (Experimental): Part A is a dose-escalation, open-label study, administering 3 doses of AdVEGF-All6A+ to n=9 individuals, with n=3 each at 10^8, 10^9, and 10^10 particle units. The purpose of Part A is to determine the highest tolerable dose. Group 1 will receive 10^9 particle units.
  Interventions: Biological: AdVEGF-All6A+
- Part A, Group 3 - 10^10 pu (Experimental): Part A is a dose-escalation, open-label study, administering 3 doses of AdVEGF-All6A+ to n=9 individuals, with n=3 each at 10^8, 10^9, and 10^10 particle units. The purpose of Part A is to determine the highest tolerable dose. Group 1 will receive 10^10 particle units.
  Interventions: Biological: AdVEGF-All6A+
- Part B, Group 1 - AdVEGF-All6A+ (Experimental): Part B (n=32 subjects) is a randomized, double blind, placebo-controlled study that will compare the AdVEGF-All6A+ vector (n=24) to a placebo, AdNull (n=8). Group 1 will receive AdVEGF-All6A+ at the highest tolerable dose determined in Part A.
  Interventions: Biological: AdVEGF-All6A+
- Part B, Group 2 - AdNull placebo (Experimental): Part B (n=32 subjects) is a randomized, double blind, placebo-controlled study that will compare the AdVEGF-All6A+ vector (n=24) to a placebo, AdNull (n=8). Group 2 will receive AdNull, the placebo vector.
  Interventions: Biological: AdNull

INTERVENTIONS:
Biological: AdVEGF-All6A+ — We will administer AdVEGF-All6A+, an adenovirus vector carrying the genetic material for human vascular endothelial growth factor to the ischemic myocardium of individuals with diffuse coronary artery disease.
  Arms: Part A, Group 1 - 10^8 pu; Part A, Group 2 - 10^9 pu; Part A, Group 3 - 10^10 pu; Part B, Group 1 - AdVEGF-All6A+
Biological: AdNull — AdNull is an adenovirus vector identical to AdVEGF-All6A+, except that it does not encode for a transgene.
  Arms: Part B, Group 2 - AdNull placebo

SUMMARY:
The proposed Phase I/II clinical trial will be used to determine the safety and toxicity of direct administration of the vector AdVEGF-All6A+ to the ischemic myocardium and to generate preliminary evidence regarding whether direct administration of AdVEGF-All6A+ to the ischemic myocardium will induce growth of collateral blood vessels and improve cardiac function. This is a three-part, multinational/multi-center, placebo controlled study.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the predominant cause of heart failure, a major cause of death and disability throughout the world. Although prognosis of patients with CAD has been greatly improved by advances in cardiovascular treatment, it is still the first cause of death in the USA. Treatment options for CAD include diet, exercise, medication, balloon angioplasty with or without stenting, atherectomy and bypass surgery. For many patients, however, the disease is diffuse and stenting or bypass surgery is not an option. A new strategy to treat these patients is to use gene therapy to induce new networks of new blood vessels to bypass the arterial system that is blocked, thus providing circulation to deliver oxygen needed by the tissue. By administering a gene coding for vascular endothelial growth factor (VEGF) to the myocardium, new networks of blood vessels can be created using the genetic material for VEGF. In experimental animal studies, VEGF is effective at treating ischemia of organs and is safe. The most direct method of transferring genes to myocardium is by injection under direct vision during a minimally invasive thoracic surgery. For the present study, the VEGF gene will be delivered to the myocardium using a modified adenovirus (Ad) as a carrier. The study is designed to test the safety and efficacy of AdVEGF-All6A+.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 90
* Demonstrable reversible left ventricular ischemia in viable myocardium as assessed by ST segment/T wave abnormalities detected by exercise testing with 99mTc-sestamibi single-photon emission computed tomography (SPECT) prior to and following the exercise test
* Individuals who have coronary artery disease (CAD) but have angina refractory to medical therapy
* Individuals who experience angina class II-IV as defined by the Canadian Cardiovascular Society
* Individuals who have had a coronary angiogram in the prior 6 months demonstrating diffuse coronary artery disease and are not considered to be eligible for coronary artery bypass surgery, stents, or angioplasty, because of the lack of suitable target lesions
* Individuals must be medically capable of undergoing open thoracotomy
* Individuals must have neutralizing anti-adenovirus serotype 5 titer ≤160; this criteria is based on the knowledge that some individuals have high anti Ad5 neutralizing antibody titer which may limit efficacy
* Hematocrit >30%
* WBC <10,000
* Normal prothrombin, partial thromboplastin time (excluding IV heparin therapy)
* Normal liver-related serum parameters
* Glomerular filtration rate (GFR) > 30 ml/min
* No evidence of active infection of any types, including adenovirus, hepatitis virus (A, B or C) or human immunodeficiency virus
* No evidence of central nervous system, major psychiatric, musculoskeletal or immune disorder
* No allergy to the vehicle used to suspend the virus or contrast materials used in radiographic procedures
* Fertile or infertile individuals; it will be recommended that fertile individuals utilize barrier birth control measures to prevent pregnancy during and for 2 months following the administration of the vector
* Individuals not receiving experimental medications or participating in another experimental protocol for at least 4 weeks prior to entry to the study.
* Individuals must be able to exercise for at least 90 seconds but no more than 15 min on a modified Bruce protocol exercise treadmill test while exhibiting angina with concurrent 1 mm horizontal or downsloping ST-segment depression
* The study individual must be able to undergo the procedures in the protocol
* Willingness to participate in the study
* Capable of providing informed consent

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria will be unable to participate in the protocol
* Individuals in whom participation in the study would compromise the normal care and expected progression of their disease
* Individuals receiving corticosteroids or other immunosuppressive medications
* Individuals with uncontrolled diabetes
* Diabetic individuals with significantly abnormal ophthalmologic exam (moderate or greater disease severity)
* Individuals with hypercholesterolemia (LDL above 190 mg/dl or total cholesterol above 240 mg/dl)
* Body mass index >35
* Recent (<6 wk) cerebral vascular accident
* Recent (<6 wk) transmural myocardial infarction
* Evidence of infection defined by elevated white blood cell (WBC) count, temperature >38.5ºC, infiltrate on chest x-ray
* Unable to undergo cardiac MRI with gadolinium contrast
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) values 2.5 greater than normal limits
* Prior cardiac transplantation
* Electrocardiograph abnormalities that would interfere with ST-segment analysis
* Untreated malignant ventricular arrhythmia
* Valvular heart disease requiring surgical intervention
* Preoperative congestive heart failure (New York Heart Association Function Class III or IV or ejection fraction (EF) <25%
* Uncontrollable asthma or chronic obstructive pulmonary disease (COPD)
* Greater than first degree heart block or sinus node dysfunction without a functional pacemaker
* Systolic blood pressure less than 90 mmHg
* Known hypersensitivity to adenosine
* Pregnancy or currently lactating
* Prior participation in cardiac gene and/or cardiac cell therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Time to 1 mm ST depression during exercise-stress testing | 3 mos (Part A); 6 mos (Part B)
  Collect the times during the stress-test

SECONDARY OUTCOMES:
Exercise-stress echocardiogram | Twice before vector administration at -30 days and -15 days (± 5 days), and will be repeated at day 90 post-vector for Part A and day 90 and 180 post-vector for Part B
  To assess segmental wall motion in treated territories
Angina | Twice pre-vector administration at -30 days and -15 days, and repeated at 30 and 90 days post-vector for Part A and at 30, 90 and 180 days post-vector for Part B
  measured by the Canadian Cardiovascular Society Functional Classification of Angina Pectoris
Cardiac MRI +/- adenosine stress | Once pre-vector and repeated at 90 days post vector for Part A, and 180 days post-vector for Part B
  To assess segmental wall motion and perfusion in treated territories

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No